CLINICAL TRIAL: NCT02123940
Title: Treatment Strategy in Patients With High-risk of Postextubation Distress in ICU Based on a Lung Ultrasound Score Versus Standard Strategy
Acronym: WIN IN WEAN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Pitié-Salpêtrière Hospital (Other); University Hospital, Grenoble (Other); Hospices Civils de Lyon (Other); Centre Hospitalier Universitaire de Saint Etienne (Other); University Hospital, Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0187; 2013-A01458-37
Record Dates: First submitted 2014-04-11; First posted 2014-04-28 (Estimated); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Adult Patients Ventilated More Than 48 h
Keywords: Weaning from mechanical ventilation; Lung ultrasound; Nasal humidified high flow therapy; Weaning failure; Postextubation distress

ARMS (2):
- nasal humidified high flow therapy (Experimental): Prospective randomized clinical multicentric study on ICU comparing a treatment strategy (nasal humidified high flow therapy and Noninvasive Ventilation) in patients with high-risk of postextubation distress in ICU based on a Lung Ultrasound Score VERSUS standard strategy
  Interventions: Device: lung ultrasound score
- standard strategy (Other): Prospective randomized clinical multicentric study on ICU comparing a treatment strategy (nasal humidified high flow therapy and Noninvasive Ventilation) in patients with high-risk of postextubation distress in ICU based on a Lung Ultrasound Score VERSUS standard strategy
  Interventions: Device: lung ultrasound score

INTERVENTIONS:
Device: lung ultrasound score — Prospective randomized clinical multicentric study on ICU comparing a treatment strategy (nasal humidified high flow therapy and Noninvasive Ventilation) in patients with high-risk of postextubation distress in ICU based on a Lung Ultrasound Score VERSUS standard strategy

SUMMARY:
Prospective, randomized clinical multicentric study in ICU during weaning from mechanical ventilation.

DETAILED DESCRIPTION:
Prospective randomized clinical multicentric study on ICU comparing a treatment strategy (nasal humidified high flow therapy and Noninvasive Ventilation) in patients with high-risk of postextubation distress in ICU based on a Lung Ultrasound Score VERSUS standard strategy

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ventilated more than 48 h
* Stable respiratory and hemodynamic conditions for SBT
* Consent of patients
* Arterial line

Exclusion Criteria:

* severe COBP
* Laryngeal dyspnea
* Tracheostomy
* Arrhythmia
* No echogenicity
* Paraplegia >T8

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 483 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2018-08-25 (Actual); Study Completion 2018-08-25 (Actual)

PRIMARY OUTCOMES:
Incidence of postextubation distress | during 48 hour (at day 1)
  postextubation period requiring a ventilatory support (reintubation or curative Noninvasive ventilation).

SECONDARY OUTCOMES:
Number of ventilator-free-days | at day 1 (after extubation)
Length of stay in ICU | at day 1
Mortality in ICU | at day 1
Extubation failure | at day 7
  Extubation failure within the 7 days following planned extubation

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien PERBET, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France